CLINICAL TRIAL: NCT01612260
Title: Shensong Yangxin Capsule in the Treatment of Mild to Moderate Systolic Heart Failure Complicated With Ventricular Premature Beat: A Randomize, Double Blind, Placebo-controlled Multicenter Clinical Trial
Brief Title: Shensong Yangxin Capsule in the Treatment of Heart Failure Complicated With Ventricular Premature Beat
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cong-xin Huang (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Fudan University (Other); Shanghai Changzheng Hospital (Other); Nanjing Medical University (Other); Third Military Medical University (Other)
Responsible Party: Sponsor-Investigator, Cong-xin Huang, professor, Wuhan University
Organization: Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: yl-yxb06-lcsyfa-201201; 2012CB518600（2012CB518606） (Other Grant/Funding Number: National Basic Research Program of China（973 Program）)
Record Dates: First submitted 2012-05-24; First posted 2012-06-05 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Heart Failure; Ventricular Premature Complex
Keywords: heart failure; ventricular premature complex; Shensong Yangxin capsule
MeSH Terms: conditions — Heart Failure; Ventricular Premature Complexes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shensong Yangxin capsule (Experimental): Shensong Yangxin capsule 4 granules t.i.d. po for 12weeks
  Interventions: Drug: Shensong Yangxin capsule
- placebo Capsule (Placebo Comparator): placebo Capsule 4 granules t.i.d. po for 12weeks
  Interventions: Drug: placebo Capsule

INTERVENTIONS:
Drug: Shensong Yangxin capsule — ShenSongYangXin Capsule 4 granules t.i.d. po for 12weeks
  Arms: Shensong Yangxin capsule
Drug: placebo Capsule — 4 granules t.i.d. po for 12 weeks
  Arms: placebo Capsule

SUMMARY:
The purpose of this study is to assess the effects of Chinese medicine Shensong Yangxin capsule for the chronic cardiac dysfunction complicated with ventricular premature beats.

DETAILED DESCRIPTION:
Premature ventricular contractions is one of the most common arrhythmia in the patients with structural heart disease and heart failure, which is not only has the high incidence but also has a high predictive value of sudden death. The purpose of the study is to assess the effects of Chinese medicine Shensong Yangxin capsule for the chronic cardiac dysfunction complicated with ventricular premature beats, which based on the numbers of premature ventricular contractions in 24-hour ambulatory electrocardiogram (ECG) as the main endpoint of the study. Secondary endpoints are evaluation of the Shensong Yangxin capsule on cardiac function and quality of life. This study is a randomized, double-blind, placebo controlled, multi-center trial. Chronic heart failure patients(cardiac function is Class II-III) associated with premature ventricular contractions (premature number 720-10000 / 24h), who received standardized treatment for heart failure at least three months, were involved in the study. Patients were randomly assigned into Shensong Yangxin capsule group or placebo group, with the capsule administration of 4 granules t.i.d.for 12 weeks. 24-hour ambulatory ECG, echocardiography and evaluation of heart function were observed at baseline and 12 weeks after the intervention. The primary outcomes are the numbers of premature ventricular contractions in 24-hour ambulatory ECG, and the secondary outcomes are New York Heart Association (NYHA) classification, NT-proBNP, left ventricular ejection fraction (LVEF) and left ventricular end-diastolic dimension (LVEDD, 6 minute walking test and Minnesota living with heart failure questionnaire (MLHFQ).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiac function NYHA II~III, Left ventricular ejection fraction (LVEF) 35%~50% tested by Modified Simpson, has a stable hemodynamics and no need to deliver treatment through vein
* To be treated by standard treatment of heart failure at least 3 months with a stable dosage already
* Ventricular premature beats: 720-10000 beats/24 hours
* Heart failure caused by ischemic heart disease, or dilated cardiomyopathy

Exclusion Criteria:

* Subject to be expected to alive no more than 6 months
* Subject suffered from acute coronary syndrome in last three months (Acute myocardial infarction of ST segment elevation and non ST segment elevation, unstable angina
* To be complicated with persistent atrial fibrillation, atrioventricular conduction block (II degree of Type II or III degree), or acute myocarditis
* To be complicated with ventricular fibrillation, torsion type ventricular heartbeat rate, sustained ventricular tachycardia, or non sustained ventricular tachycardia with rapid ventricular rate and hemodynamic disorders
* Sinus heart rate less than 45 beats/minutes and needs to receive the pacemaker or has received pacemaker, or with abnormal sinus node function
* The hypertension, diabetes difficult to be controlled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
numbers of the Premature ventricular contractions during 24-hour ambulatory ECG | 3 months

SECONDARY OUTCOMES:
NYHA classification | 3 months
LVEF | 3 months
NT-proBNP | 3 months
Minnesota living with heart failure questionnaire (MLHFQ) | 3 months
6 minute walking test | 3 months
LVEDD | 3 months

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Anzhen Hospital, Capital University of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Freindship Hospital, Beijing, Beijing Municipality
  - Chongqing Zhongshan Hospital, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The first hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Enshi Autonomous Region Central Hospital, Enshi, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - General Hospital of Dongfeng Motor Corporation, Shiyan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First College of Clinical Medical Science, China Three Gorges University, Yichang, Hubei
  - First hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital,The Affiliated hospital of Nanjing University Medical school, Nanjing, Jiangsu
  - The General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Traffic hospitals of Shandong Province, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Westchinahospital,Sichuanuniversity, Chengdu, Sichuan

REFERENCES:
- [Derived] Wang X, Hu D, Dang S, Huang H, Huang CX, Yuan MJ, Tang YH, Zheng QS, Yin F, Zhang S, Zhang BL, Gao RL; Efficacy and Safety of Shensong Yangxin Capsules for Frequent VPCs in Congestive Heart Failure Study Group. Effects of Traditional Chinese Medicine Shensong Yangxin Capsules on Heart Rhythm and Function in Congestive Heart Failure Patients with Frequent Ventricular Premature Complexes: A Randomized, Double-blind, Multicenter Clinical Trial. Chin Med J (Engl). 2017 Jul 20;130(14):1639-1647. doi: 10.4103/0366-6999.209906. PMID 28685712